CLINICAL TRIAL: NCT04284358
Title: Comparison of Workshop Delivery Methods on Youth Soccer Coaches' Ability to and Self-efficacy in Identifying Exercise Errors of a Soccer Neuromuscular Training Warm-up
Brief Title: Does Peer to Peer Learning Facilitated by an iPad Application Help Coaches Learn a Neuromuscular Training Warmup?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport Injury Prevention Research Centre (Other)
Responsible Party: Principal Investigator, Kati Pasanen, PT MSc PhD, Assistant Professor, Sport Injury Prevention Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soccer NMT
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Sport Injury
Keywords: Neuromuscular Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into the control or intervention NMT warm-up workshop. The integration of peer to peer learning technology into the workshop is the intervention aspect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Instruction workshop (No Intervention): Standard instruction neuromuscular training warm-up workshop. Participants will learn of the exercises with a traditional instructor demonstration and verbal explanation and then attempt it themselves.
- Technology Integrated Instruction workshop (Experimental): Technology integrated instruction neuromuscular training warm-up workshop. Participants will learn of the exercises with a traditional instructor demonstration and verbal explanation and. Participants will then attempt the exercise and assess their execution via a video on a peer learning tablet application.
  Interventions: Other: Technology integrated instruction neuromuscular training warm-up workshop

INTERVENTIONS:
Other: Technology integrated instruction neuromuscular training warm-up workshop — Participants will learn of the exercises with a traditional instructor demonstration and verbal explanation. Participants will then attempt the exercise and assess their execution via a video on a peer learning tablet application. This occurs for every exercise and occurs in pairs in which participants can discuss and evaluate an exercise by an exercise's key execution components.
  Arms: Technology Integrated Instruction workshop

SUMMARY:
Purpose: To compare standard or technology integrated workshop delivery on coaches' measured ability to and confidence in recognizing for errors for key components of exercises in a soccer neuromuscular training (NMT) warm-up. Research in this area is needed to measure how effective NMT warm-up workshops are on educating coaches and if technology integration into the workshop improves their understanding as these measures are unknown to date.

Background: Injury prevention strategies such as using a NMT warm-up has been successful in reducing injuries (Emery, Roy, Whittaker, Nettel-Aguirre, & van Mechelen, 2015). NMT warm-up workshops are provided to educate coaches however there are adoption issues for the coaches (van Reijen, Vriend, van Mechelen, Finch, & Verhagen, 2016). An effective workshop is designed to enhance a coaches' self-efficacy and have a practical portion to work through the exercises (Emery, 2015; Steffen et al., 2013). iPad applications such as the Move Improve application are utilized to enhance peer to peer learning and provide feedback for the subject performing the exercise.

Research Plan: A randomized controlled trial (RCT) will be performed with clubs from the Calgary Minor Soccer Association (CMSA). Coaches from the recruited clubs will be randomized to attend one of two types of workshops : 1) intervention group (technology integrated coach NMT warm-up workshop) and 2) control group (standard NMT warm-up workshop.The control workshop is a two-hour workshops that includes an information period, on field instruction and partnered practice for all soccer NMT exercises. The technology-based workshop which is a two-hour workshop that includes on field exercise instruction and then partnered practice with use of the Move Improve mobile application for all soccer NMT exercises. All coaches (n=100; 50 per group) prior to the workshop commencing interested participants with be asked to fill out the consent form, the soccer NMT demographic information form and the Soccer NMT warm-up exercise self-efficacy questionnaire. Following the workshop, coaches will be asked to complete Soccer NMT warm-up exercise self-efficacy questionnaire again and the soccer NMT warm-up exercise test.

DETAILED DESCRIPTION:
Study Design A cluster randomized controlled trial (RCT) was conducted within the Calgary Minor Soccer Association (CMSA) in 2019 to evaluate how integration of peer to peer (P2P) learning with technology into a soccer NMT warm-up workshop influences coaches' ability and confidence to identify exercise errors. Soccer coaches within each recruited club were randomly educated with a soccer NMT warm-up workshop with or without peer to peer learning technology. Coaches completed a video-based test and self-efficacy scale on their ability to recognize NMT exercise errors.

Participants and Randomization The study population included CMSA youth soccer coaches during the 2019/2020 indoor soccer season. The forty soccer clubs of the CMSA received a study information flyer by e-mail from the CMSA administration staff. Six of the soccer clubs agreed to host soccer NMT warm-up workshops at their club houses for a total of 89 youth soccer coaches in attendance.

Coaches from the recruited clubs were randomized to attend one of two types of workshops; the intervention workshop with technology integrated instruction of the soccer NMT warm-up or the control workshop with standard in person instruction of the soccer NMT warm-up. A stratified by soccer club and block randomized by two (for each type of workshop) computer generated randomized allocation sequence was used to determined which workshop the coaches receive within each club. The randomized allocation sequence was generated prior to the study commencing by the investigator. As clubs were recruited and workshops were scheduled, assignment of the interventions were applied by the investigator to workshop facilitators prior to workshop delivery.

Procedures Soccer NMT Warm-up Program The soccer NMT warm-up program is a modified version of a NMT warm-up program developed by Finnish researchers for floorball and soccer by Pasanen et al. (2008). This program is also a slightly modified version of the presently used SHRed Injuries NMT warm-up program. The current soccer NMT program consists of nine, level one exercises divided into four categories: aerobic, agility, strength, and balance where most exercises have the option to increase the difficultly as shown by the level two options.

Peer to Peer Learning Tablet Application The P2P learning tablet-based application is an application used to facilitate the comprehension and execution of various movement patterns. This is the technology that will be used in the intervention workshop. For each movement pattern or exercise, the application requires two individuals to partner up where one is the subject performing the exercise in the video recorded (video not to be stored on the application or device) and the other individual records the video. Prior to recording any video, the partners observe a correct exercise demonstration video and a list of key criteria or key components for every exercise that has to be met in order for the exercise to be performed correctly. One person in the partnership is filmed performing the exercise. The subject and their partner are then able to view the video, evaluate it and discuss if the subject was able to perform each component correctly, incorrectly or partially correct. The partners then switch roles. Application users are then able to improve their execution and understanding of the exercise by evaluating themselves and their partner through the application.

Data Collection Two types of soccer NMT workshops were offered. The intervention group received the technology integrated instruction workshop which was a two-hour workshop that included information on injury risks and NMT, on field exercise instruction with instruction on how to use the P2P learning tablet application followed by partnered practice with use of the application for all soccer NMT warm-up exercises. The control group received the standard in person instruction workshop (without technology). This was a two-hour workshop that included information on injury risks and NMT, on field instruction and partnered practice for all soccer NMT warm-up exercises. A pilot intervention workshop occurred (n=3) to optimize the workshop's delivery. All coaches were provided with copies of the soccer NMT warm-up program with pictures of all the exercises with required repetitions and supplementary materials.

Data was collected at the beginning and the end of the soccer NMT warm-up workshops. At the beginning, participants consented, provided basic demographic information and completed the soccer NMT warm-up exercise self-efficacy questionnaire. Following the completion of the workshop, participants completed the soccer NMT warm-up exercise self-efficacy questionnaire again, and the soccer NMT warm-up exercise test.

Measures The outcomes of this study are assessing the change in coaches' self-efficacy and ability to identify exercise errors. In addition, basic demographic information was collected to allow to describe the sample and use advanced statistical analysis methods.

Self- Efficacy Scale Soccer NMT warm-up exercise self-efficacy questionnaire was developed as a nine item 7 point Likert scale. This scale was developed to assess coaches (in lay terms) confidence to recognize incorrect exercise execution for each exercise. Coaches were presented with the stem question "How confident are you in your ability to see mistakes when as athlete performs the exercise…" followed by the name of each of the evaluated level one exercises within the Soccer NMT Warm-up program. The Likert scale ranged from Not Confident at All to Somewhat Confident to Completely Confident.

Coaches were asked to complete the mobile administered scale at the beginning of the workshop prior to being introduced to the exercises. To eliminate any confusion about exercises that have multiple names for example, coaches watched a short video introducing what the exercises are and the names for them being used in the soccer NMT warm-up. Coaches were asked again to complete the scale at the end of the workshop after learning the exercises. At both time points, the mean of the nine items was taken to score the scale. The change in coaches' self-efficacy was calculated by taking the difference between time points for each participant.

Video-based Exercise Test Soccer NMT warm-up exercise test was created to provide an objective measure of coaches' ability to recognize incorrect exercise execution of the soccer NMT warm-up exercises. 16 multiple choice questions with four response options were developed. For each question, participants needed to watch a video of an athlete performing one execution error for one of nine level one exercises. The participants were asked to identify which component of the exercise is being performed incorrectly by selecting the false response option. The response options for these exercises were modified from the performance criteria components of the SHRed Basketball Warm-up Observational Tool. The tool breaks down an exercise to its essential components to assess fidelity, whether an athlete is performing an exercise correctly by all of its components. The responses stem from the tool as many of the basketball and soccer NMT warm-up exercises are the same and the tool was also used to assess exercise fidelity through video analysis.

An example of a question is as follows:

A total of 16 points was allotted for this test, one per correctly identified error. One to two points per exercise was allotted for injury prevention focuses (11 points) and one to two per exercise (five points) was allotted for the key execution components that are not explicitly injury prevention focused.

Descriptive Statistics Demographic Information Participants who did not complete the necessary forms fully or correctly were identified and removed. Demographic participant information was screened to identify errors, missing data and/ or outliers. Data that could be collected by following up with the participant was added. Missing demographic info was not imputed. Soccer NMT warm-up exercise self-efficacy data with missing values were imputed with the mean of the remaining items within the scale for when that participant's questionnaire had at least half of the items completed. Internal consistency (Cronbach's alpha) was calculated for the soccer NMT warm-up exercise self-efficacy questionnaire at both time points. Intraclass correlation was calculated to estimate the degree of clustering between soccer clubs for all outcomes. Data were analyzed using STATA 15.1 software. Data was analyzed and summarized with descriptive statistics based on the workshop the coach attended such as sample. Data that could be reported through measures of central tendency underwent distribution assessment and were reported appropriately (means and standard deviations or medians with ranges) such as soccer NMT warm-up exercise test scores, the change in mean soccer NMT warm-up exercise self-efficacy scores, age and number of years coaching. Remaining variables were reported as a dichotomous yes or no such as sex, previous injury prevention program use, volunteer coach status, and personal training experience.

Exploratory Objectives Descriptive statistics by proportions were used to depict the percentage of correctly identified errors by soccer NMT warm-up exercise test injury prevention test focuses.

Multivariable Analysis Primary Objectives Multiple linear regression analyses were used to determine if an association existed between soccer NMT warm-up workshop attended (control vs intervention workshop) and outcomes soccer NMT warm-up exercise test scores (score out of 16) and the change in mean soccer NMT warm-up exercise self-efficacy scores (within the 7 point Likert scale). These outcome variables are being assessed as continuous variables. Other covariate variables to be included in both regression analyses were age (years), sex (male/ female), number of years coaching soccer (years), previous use of any injury prevention program (yes/no), being volunteer coach (yes/no), soccer NMT warm-up exercise test scores or the change in mean soccer NMT warm-up exercise self-efficacy if they were not the outcome of that analysis and, were adjusted for any effects of clustering by club. All covariates in these analyses were able to be potential modifiers and/or confounders in the regression analyses, which were assessed using a backwards elimination process. Results were reported as estimations of mean test scores and change in mean self-efficacy scores for the final models from the linear regression analyses.

Statistical significance level for all analysis was set at 5% (alpha=0.05). The outcomes of this study are novel thus sample size is unable to be determined by calculation. However, an estimate of 10 participants per beta coefficient included in the model was used to estimate a feasible sample size of n=100 (50 per group) as per statistician recommendation. In addition, based on previous studies conducted in Calgary through the Sport Injury Prevention Research Centre, typically the most amount of coaches to have participated in CMSA soccer related studies is 60 coaches.

ELIGIBILITY:
Inclusion Criteria:

* Youth Soccer Coaches in the Calgary Minor Soccer Association

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Soccer neuromuscular training warm-up exercise test | immediately after the workshop (control or intervention)
  A multiple choice test with video based questions where participants are asked to identify the exercise error in the video.
Change in soccer neuromuscular training warm-up exercise self-efficacy by scale | immediately after and just before (10-15 min) the workshop (control or intervention)
  A confidence scale assessing participant's confidence in their ability to identify exercise errors for every exercise in the warm-up. On a 0 to 7 point Likert scale where the mean higher score indicates more confidence or a better outcome. The change in self-efficacy is calculated by taking the difference in mean scores between time points.

CONTACTS AND LOCATIONS:
Overall Officials: Kati Pasanen, PhD, Principal Investigator — Sport Injury Prevention Research Centre
Locations (1):
- Sport Injury Prevention Research Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emery C, Tyreman H. Sport participation, sport injury, risk factors and sport safety practices in Calgary and area junior high schools. Paediatr Child Health. 2009 Sep;14(7):439-44. doi: 10.1093/pch/14.7.439. PMID 20808471
- [Background] Emery CA, Roy TO, Whittaker JL, Nettel-Aguirre A, van Mechelen W. Neuromuscular training injury prevention strategies in youth sport: a systematic review and meta-analysis. Br J Sports Med. 2015 Jul;49(13):865-70. doi: 10.1136/bjsports-2015-094639. PMID 26084526
- [Background] Steffen K, Meeuwisse WH, Romiti M, Kang J, McKay C, Bizzini M, Dvorak J, Finch C, Myklebust G, Emery CA. Evaluation of how different implementation strategies of an injury prevention programme (FIFA 11+) impact team adherence and injury risk in Canadian female youth football players: a cluster-randomised trial. Br J Sports Med. 2013 May;47(8):480-7. doi: 10.1136/bjsports-2012-091887. Epub 2013 Mar 13. PMID 23486935
- [Background] van Reijen M, Vriend I, van Mechelen W, Finch CF, Verhagen EA. Compliance with Sport Injury Prevention Interventions in Randomised Controlled Trials: A Systematic Review. Sports Med. 2016 Aug;46(8):1125-39. doi: 10.1007/s40279-016-0470-8. PMID 26869058